CLINICAL TRIAL: NCT03859336
Title: High-Frequency Transdermal Neuromodulation to Decrease Anxiety and Improve Sleep in Autism Spectrum Disorder (ASD)
Brief Title: High-Frequency Transdermal Neuromodulation to Decrease Anxiety and Improve Sleep in ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Richard Frye, MD, PhD, Chief of Neurodevelopmental Disorders at Barrow Neurological Institute, Phoenix Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TENS_ASD
Record Dates: First submitted 2019-02-21; First posted 2019-03-01 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Anxiety; Sleep Issues
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective 3 day open-label device trial across all subjects, with 1 day single-blinded sham pre- and post-treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transdermal Neuromodulation Stimulation (Experimental): Day 1 of Transdermal Neuromodulation Stimulation (TENS) is a one-day sham stimulation, consisting of: 30 seconds of sensation in which amplitude is increased up to the threshold of salient sensation, followed by 19 minutes of no stimulation (device is turned off), followed by 30 more seconds of salient stimulation. Day 1 is used to exclude those who cannot tolerate study procedures and placebo responders; it will also serve as baseline for anxiety measures. TENS treatment begins one day after sham, and lasts 3 days with 20 minutes of stimulation per day. One day following open label treatment all participants will once again receive sham stimulation following the same procedures utilized at Day 1.
  Treatment amplitude is adjusted for each participant, in which the stimulation will be administered just below the participant's sensation threshold. Amplitude from the TENS device does not exceed 20mA. Frequency will be at 300hz.
  Interventions: Device: Transdermal Neuromodulation Stimulation

INTERVENTIONS:
Device: Transdermal Neuromodulation Stimulation — The TEN device administers a tuned high frequency electrical stimulation delivered to the cervical plexus (C2-C4) on the back of the neck for 20 minutes. This stimulation will activate common trigeminovagal pathways modulating noradrenergic signaling to attenuate sympathetic activity. This stimulation can subsequently regulate the activity of several deep-brain nuclei within the ascending reticular activating system (RAS). Nuclei in the RAS regulate powerful neuromodulators like norepinephrine (NE), acetylcholine (ACh), and serotonin (5-HT). The investigators will examine whether this modulation from TENS will decrease anxiety and improve sleep quality in the study participants.

SUMMARY:
The objective of this study is to investigate the feasibility of cervical TEN stimulation (TENS) delivered to the back of the neck to decrease anxiety and sleep issues in young adults with Autism Spectrum Disorder (ASD). The specific aim is to determine the effect of TENS, delivered over 3 daily sessions, on anxiety and sleep quality in young adults with ASD, as compared to sham and baseline. The investigator will enroll up to 10 young adults, aged 10 to 25 years of age with confirmed ASD and measureable anxiety and sleep disturbance symptoms, and participation will last 3 weeks.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a heterogeneous neurodevelopmental disorder with life-long consequences that affects children during critical times in their development. ASD is associated with co-occurring problems such as anxiety and sleep disturbances. New approaches to managing stress, anxiety, and sleep quality would greatly enhance the quality of life and activities of daily living for children with ASD as they transition to adulthood and age out of services. Based on strong evidence from typically developing individuals, the technology for transdermal electrical neuromodulation (TEN) of the cranial nerves has shown to be a safe, effective, comfortable, and non-pharmacological therapy to modulate the central nervous system decreasing anxiety and enhancing sleep quality to improve the quality of life for people with ASD.

The therapy applies tuned, high-frequency TEN to the back of the neck which activates the brainstem modulating noradrenergic signaling shown to decrease anxiety in healthy adults. The low-amplitude of the stimulation means that it is painless and comfortable. Furthermore, the technology is being evaluated for improving sleep quality. The mechanism of these effects are well established in the neurophysiology literature, but modulating these brainstem areas is only now possible non-invasively with the technology. Participants entered into the trial wil have anxiety and sleep issues that are known to be associated with ASD. The investigators hypothesize that cervical TEN will decrease anxiety and improve sleep quality in a population with high-functioning ASD who are transitioning into adulthood.

The investigators will study 10 young adults, between the ages of 10 years to 25 years, with confirmed ASD and anxiety and sleep quality issues. All participants will be enrolled in the study for approximately 2 weeks. During the first week, participants will undergo 5 consecutive days of stimulation. On Visit 1, all participants will receive sham stimulation, which will be used to exclude placebo responders and those who cannot tolerate study procedures, and determine the maximum stimulation threshold for eligible participants. Additionally, the visit will serve as the baseline day to collect measures of anxiety. The primary physiological anxiety measures include galvanic skin response (GSR) and heart rate variability (HRV). Secondary measures will include data from behavioral surveys, and cortisol and amylase analyses from passive drool samples. Participants will report baseline sleep habits in the form of a questionnaire.

If all eligibility criteria are met, participants will return for 3 consecutive days of open label TEN stimulation treatment. Anxiety measures will be collected at each visit. On the fifth consecutive day, participants will once again receive sham stimulation in order to determine the impact of the open label treatment. Participation will conclude with a one day phone follow-up visit one week from the last treatment day. Caregivers will report participant sleep quality and any adverse effects or changes.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 10 - 25 years old
* IQ > 80, to be evaluated during the screening visit using the Kaufman Brief Intelligence Test (KBIT)
* Self-reported complaints about anxiety and/or sleep issues
* Screen for Child Anxiety Related Disorders (SCARED) - Parent Form, score >= 25
* Able to follow directions in English

Exclusion Criteria:

* • IQ ≤ 80, to be evaluated during the screening visit using the KBIT
* SCARED - Parent Form, Score < 25
* Has a medical implant (such as a pacemaker, cochlear implant, brain stimulation device, spinal stimulator)
* History of significant face/head injury including cranial or facial metal plate or screw implants
* Pregnant
* History of migraines or frequent headaches (more than once a week)
* Started taking anti-anxiety medications less than 3 months prior to study participation or has not been taking anti-anxiety medications consistently for at least 3 months prior to study participation
* Fainting (vaso-vagal syncope or neurocardiogenic syncope)
* Diagnosis of Raynaud's disease
* Tempromandibular joint (TMJ) disorder or other facial neuropathy
* Poor vision or hearing that is uncorrectable
* Seizures in the last 2 years
* Evidence of skin disease or skin abnormalities affecting the neck or upper back
* Upper extremity contractures

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Change in physiological response measure of heart rate variability in the time-domain as measured by the standard deviation of the normal-to-normal heart beat (SDNN) | Baseline Visit (Day 1), Treatment Visits (Days 2, 3, and 4), Sham Visit (Day 5)
  The standard deviation of the normal-to-normal heart beat (SDNN) is the time-domain based measured of heart rate variability. It is measured by calculating the standard deviation of the heart beat-to-beat time interval, which is measured in milliseconds. Anxiety reduction will be demonstrated by a reduction in the SDNN value during a stressor in response to TEN treatment, as compared to baseline.
Change in physiological response measure of heart rate variability in the frequency-domain as measured by the power of the low frequency (LF) band | Baseline Visit (Day 1), Treatment Visits (Days 2, 3, and 4), Sham Visit (Day 5)
  The low frequency (LF) component of heart rate variability (HRV) is the frequency band ranging from 0.04-0.15Hz of the waveform created by heart rate oscillations. Spectral power is calculated for this band in milliseconds squared. Anxiety reduction will be demonstrated by a reduction in the power value of the LF HRV component during a stressor in response to TEN treatment, as compared to baseline.
Change in physiological response measure of heart rate variability in the frequency-domain as measured by the power of the high frequency (HF) band | Baseline Visit (Day 1), Treatment Visits (Days 2, 3, and 4), Sham Visit (Day 5)
  The high frequency (HF) component of heart rate variability (HRV) is the frequency band ranging from 0.15-0.4Hz of the waveform created by heart rate oscillations. Spectral power is calculated for this band in milliseconds squared. Anxiety reduction will be demonstrated by a reduction in the power value of the HF HRV component during a stressor in response to TEN treatment, as compared to baseline.
Change in physiological response measure of galvanic skin response (GSR) | Baseline Visit (Day 1), Treatment Visits (Days 2, 3, and 4), Sham Visit (Day 5)
  Galvanic skin response (GSR) is an electrodermal conductance measurement that reflects the changes in sweat gland activity, which is measured in microsiemens (μS). Anxiety reduction will be analyzed through a suppression of GSR activity value during a stressor in response to TEN treatment, as compared to baseline data.

SECONDARY OUTCOMES:
Change in the Screen for Child Anxiety Related Disorders (SCARED) score | Baseline Visit (Day 1), Treatment Visits (Days 2, 3, and 4), Sham Visit (Day 5)
  The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item self-reported inventory that measures anxiety in youth with ASD. Each item rates the severity of a symptom or behavior on a 3 point scale from 0 (Not true or Hardly Ever True) to 2 (Very True or Often True). A decrease in the total score of the 41 items, ranging from 0 to 82, will be used as a secondary measure to define a positive response.
Change in the Parent Reported Anxiety Scale (PRAS) score | Baseline Visit (Day 1), Treatment Visits (Days 2, 3, and 4), Sham Visit (Day 5)
  The Parent-rated Anxiety Scale for Autism Spectrum Disorder is a 25-item scale that measures anxiety in youth with ASD. Each item rates the severity of a behavior on a 4 point scale from 0 (None/not present) to 3 (Severe/Very frequent and a major problem). A decrease in the total score of the 25 items, ranging from 0 to 75, will be used as a secondary measure to define a positive response.
Change in amylase and cortisol levels | Baseline Visit (Day 1), Treatment Visits (Days 2, 3, and 4), Sham Visit (Day 5)
  Another secondary outcome measure for anxiety will be to quantify α-amylase and cortisol levels in the collected saliva samples, comparing post-treatment sample levels to pre-treatment within a visit. Successful anxiety reduction will be demonstrated by reduced levels of α-amylase and cortisol in the sample as compared to pre-TEN treatment levels.
Change in the Children's Sleep Habits Questionnaire (CSHQ) score | Baseline Visit (Day 1), Treatment Visits (Days 2, 3, and 4), Sham Visit (Day 5), Follow-Up (1 week following sham visit)
  The Children's Sleep Habits Questionnaire (CSHQ) is a 39-item informant-reported questionnaire that measures sleep quality in children. Each item rates the frequency of a sleeping behavior on a 3 point scale from 1 (Never/Rarely, 0-1 nights per week) to 3(Usually, 5-7 nights pers week). The questionnaire also consists of questions asking whether certain behaviors are a problem with the options of a "yes" or "no" response.
  Improved sleep quality will be determined by a decrease in scores on the CSHQ subscales and the CSHQ combined total score, ranging from 31-93.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, MD, PhD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

REFERENCES:
- [Background] Tyler WJ, Boasso AM, Mortimore HM, Silva RS, Charlesworth JD, Marlin MA, Aebersold K, Aven L, Wetmore DZ, Pal SK. Transdermal neuromodulation of noradrenergic activity suppresses psychophysiological and biochemical stress responses in humans. Sci Rep. 2015 Sep 10;5:13865. doi: 10.1038/srep13865. PMID 26353920
- [Background] Boasso AM, Mortimore H, Silva R, Aven L, Tyler, WJ. Transdermal electrical neuromodulation of the trigeminal sensory nuclear complex improves sleep quality and mood. BioRxiv. 2016 Jan 1. doi: 10.1101/043901
- [Background] Carter ME, Yizhar O, Chikahisa S, Nguyen H, Adamantidis A, Nishino S, Deisseroth K, de Lecea L. Tuning arousal with optogenetic modulation of locus coeruleus neurons. Nat Neurosci. 2010 Dec;13(12):1526-33. doi: 10.1038/nn.2682. Epub 2010 Oct 31. PMID 21037585
- [Background] van Steensel FJA, Heeman EJ. Anxiety Levels in Children with Autism Spectrum Disorder: A Meta-Analysis. J Child Fam Stud. 2017;26(7):1753-1767. doi: 10.1007/s10826-017-0687-7. Epub 2017 Mar 20. PMID 28680259
- [Background] White SW, Oswald D, Ollendick T, Scahill L. Anxiety in children and adolescents with autism spectrum disorders. Clin Psychol Rev. 2009 Apr;29(3):216-29. doi: 10.1016/j.cpr.2009.01.003. Epub 2009 Jan 25. PMID 19223098